CLINICAL TRIAL: NCT02942927
Title: Team Approach to Polypharmacy Evaluation and Reduction Randomized Controlled Trial
Brief Title: Team Approach to Polypharmacy Evaluation and Reduction
Acronym: TAPER-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); David Braley and Nancy Gordon Chair in Family Medicine (Other); RxISK (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RN293982 - 367123
Record Dates: First submitted 2016-08-22; First posted 2016-10-24 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2023-10

CONDITIONS: Multi-morbidity; Medication Therapy Management; Polypharmacy
Keywords: Polypharmacy; Multimorbidity; Randomized Control Trial; Drug Discontinuation; Patient Preference; eHealth
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI and Data analyst were blinded to allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAPER (Experimental): The intervention is medication reduction. This arm is comprised of:
  1. Medication reconciliation
  2. Identification of patient priorities for care
  3. Identification of medications that are potentially appropriate for discontinuation/dose reduction
  4. Linked pharmacist/family physician consultations with patient to discuss medication with intention to reduce
  5. Identification of medications for trial of discontinuation/dose reduction (shared decision making)
  6. Pause of medication and clinical monitoring
  Interventions: Other: Medication reduction
- Control (No Intervention): Standard of Care as wait list control. Control group will be offered intervention as part of usual clinical care at 6 months.

INTERVENTIONS:
Other: Medication reduction — Systematic approach to reduction in polypharmacy.
  Other Names: Medication discontinuation/dose reduction
  Arms: TAPER

SUMMARY:
In an aging population, most seniors suffer from multiple chronic conditions. When the number of medications taken is ≥5 (polypharmacy), the burden of taking multiple concurrent medications can do more harm than good. Seniors take an average of 7 regular medications and studies link polypharmacy with adverse effects on morbidity, function and health service use. However, it is not clear to what extent these are reversible if medication burden is reduced.

This trial will test the effects on medication numbers and patient health outcomes of an intervention to polypharmacy. This study will test a program focused on medication reduction number and dose. Prioritizing medications according to the patient's preference as reducing the dose also reduces the risk of drug side effects.

Patients, aged 70 years of age or older and are taking ≥5 medications, will randomly receive the program immediately or at 6 months. The program involves information gathering from the patient, including systematically seeking patients priorities and preferences medication review with the pharmacist and then a consultation with the family doctor. The intervention is focused on discontinuing/reducing the dose of medications where possible using a 'pause and monitor' framework to assess the need for restart. An electronic program that detects drug adverse effects and flags potentially inappropriate medications will be integrated into an electronic clinical pathway incorporating monitoring and follow up systems.

This study will examine effects on patient and health relevant outcome measures as well as qualitative research exploring patients' and clinicians' experiences of reducing medication burden. The results will be used to determine whether this system can be implemented as part of routine preventative care in primary care for older adults.

DETAILED DESCRIPTION:
Patients will be randomized 1:1 to receive the intervention at study start or delayed appointment 6 months later. Initial baseline data collection from the patient include data on demographics, medications, and illness characteristics. The patient will then attend an appointment with a pharmacist to review medications appropriate for discontinuation/dose reduction, after which the patient will meet with their family physician to discuss patient preferences for discontinuation/dose reduction. Both health care providers will have access to TaperMD, a web based program linked to evidence and tools to support reduction in polypharmacy. Follow-up research assessments will take place at one week, 3 months and 6 months (study end). Outcome assessments and a semi-structured interview will take place at the 6 month appointment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years of age or older
* Patient must have a family doctor
* Participating family doctor as most responsible provider
* Currently taking more 5 or more long-term medications
* Have not had a recent (past 12 months) comprehensive medication review
* Patient willing to try discontinuation

Exclusion Criteria:

* English language or cognitive skills inadequate to understand and respond to rating scales
* Terminal illness or other circumstance precluding 6 month study period

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 345 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Successful discontinuation (mean difference in number of medications) | Baseline, 6 months
  Difference in mean number of medications

SECONDARY OUTCOMES:
Quality of life (EQ5D-5L) | Baseline, 6 months
  EuroQol five dimensions questionnaire (EQ5D-5L)
Quality of life (SF36v2) | Baseline, 6 months
  The Short Form (36) Health Survey (SF-36-V2)
Cognition | Baseline, 6 months
  The Mini Mental Status Examination (MMSE)
Fatigue | Baseline, 6 months
  Avlund Mob-T Scale
Patient experience of pain | Baseline, 6 months
  Brief Pain Inventory (Pain interference and Pain severity sub-scales)
Patient enablement | Baseline, 6 months
  The Patient Enablement Index (PEI)
Sleep | Baseline, 6 months
  15-D Scale (Sleep Question)
Disease burden | Baseline, 6 months
  Disease Burden Survey (Bayliss et al., 2009)
Nutritional status | Baseline, 6 months
  Mini Nutritional Assessment Short-Form (MNA-SF)
Treatment burden | Baseline, 6 months
  Brief Treatment Burden Scale
Falls | Baseline, 6 months
  Total number of falls resulting in medication consultation or treatment recorded in hospital admission and primary care records, and by patient
Physical functional capacity and ability | Baseline, 6 months
  Manty structured validated interview
Physical function capacity and ability (timed-up-and-go) | Baseline, 6 months
  Timed up and go test (TUG)
Physical function capacity and ability (strength) | Baseline, 6 month
  Grip strength
Physical function capacity and ability (balance) | Baseline, 6 months
  Global Rating of Change (Balance)
Healthcare resource utilization (hospital admissions) | Baseline, 6 months
  Number of hospital admissions from administrative data and self-report; proportion of patients with at least one hospitalization
Healthcare resource utilization (ED/urgent care visits) | Baseline, 6 months
  Number of emergency department and urgent care visits from administrative data and self-report
Healthcare resource utilization (primary care visits) | baseline, 6 months
  Number of primary care visits from administrative data
Successful discontinuation or dose reduction | 6 months
  Composite variable calculate to represent mean number of medications stopped or dose reductions
Successful discontinuation or dose reduction (proportion) | 6 months
  Proportion of patients with successful discontinuations or dose reductions
Changes in medication side effects and symptoms (adverse) | 1 week, 3 month, 6 month
  Patient self-report of appearance (new or worsening) of side effects associated with medications
Changes in medication side effects and symptoms (positive) | 1 week, 3 month, 6 month
  Patient self-report of disappearance (improvement or disappearance) of side effects associated with medications
Serious adverse events | 3 months, 6 months
  Any event that requires in-patient hospitalization or prolongation of existing hospitalization, causes congenital malformation, results in persistent or significant disability or incapacity, is life-threatening or results in death (Health Canada (2011) Guidance Document for Industry - Reporting Adverse Reactions to Marketed Health Products)
Medication self-efficacy | Baseline, 6 months
  Self-efficacy for appropriate mediation use scale

OTHER OUTCOMES:
Implementation processes | baseline, 3 months, 6 months
  NoMAD survey
Pharmacists/family physician 5 best/worst aspects of intervention | 6 months
  Open ended list
Pharmacists/family physician confidence in medication discontinuation | Baseline, 6 months
  5 point Likert scale single question developed for study
Pharmacists/family physician experiences with the deprescribing process | 6 months
  Semi-structured interviews; field notes
Strengths and weaknesses of intervention | 6 months
  Open ended questions
Patient experience with deprescribing process (diary) | 6 months
  Patient diaries
Patient experience with deprescribing process (interview) | 6 months
  Semi-structured interview
Satisfaction with intervention | 6 months
  5 point Likert scale single question developed for study
Satisfaction with care around medications | Baseline, 6 months
  5 point Likert scale single question developed for study
Cost effectiveness | 6 months
  Incremental cost per Quality Adjusted Life Year (payer perspective)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Dee Mangin, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mangin D, Lamarche L, Agarwal G, Banh HL, Dore Brown N, Cassels A, Colwill K, Dolovich L, Farrell B, Garrison S, Gillett J, Griffith LE, Holbrook A, Jurcic-Vrataric J, McCormack J, O'Reilly D, Raina P, Richardson J, Risdon C, Savelli M, Sherifali D, Siu H, Tarride JE, Trimble J, Ali A, Freeman K, Langevin J, Parascandalo J, Templeton JA, Dragos S, Borhan S, Thabane L. Team approach to polypharmacy evaluation and reduction: study protocol for a randomized controlled trial. Trials. 2021 Oct 26;22(1):746. doi: 10.1186/s13063-021-05685-9. PMID 34702336